CLINICAL TRIAL: NCT06020534
Title: Safety and Efficacy of Kidney Transplantation in Patients With Aortoiliac Stenosis
Brief Title: Aortoiliac Stenosis in Kidney Transplantation
Acronym: TASC
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Yitian Fang, MD, Principal Investigator, Erasmus Medical Center
Other Study IDs: KT TASC
Record Dates: First submitted 2023-08-24; First posted 2023-08-31 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Aorto-Iliac Arterial Stenosis; Peripheral Arterial Disease; Kidney Transplant Failure
Keywords: aortoiliac arterial stenosis; peripheral arterial disease; kidney transplantation; outcomes
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No-stenosis group: Patients who had no pre-existing aortoiliac stenosis before kidney transplantation.
- TASC A/B stenosis: Patients who had TASC A or B aortoiliac stenosis before kidney transplantation.
- TASC C/D stenosis: Patients who had TASC C or D aortoiliac stenosis before kidney transplantation.

SUMMARY:
The impact of aortoiliac stenosis on kidney transplant patients remains unclear. This study aims to investigate the safety and efficacy of kidney transplantation in patients with aortoiliac stenosis.

DETAILED DESCRIPTION:
Kidney transplantation is the optimal treatment for end-stage renal disease (ESRD). Unfortunately, not all ESRD patients are eligible for kidney transplantation. Aortoiliac stenosis, an increasingly common type of peripheral arterial disease in ESRD patients, is considered as relative contra-indication for kidney transplantation. There are several reasons for concern, such as the complexity of the vascular anastomosis and inferior life expectancy. Consequently, it is still debated whether patients with aortoiliac stenosis would benefit from kidney transplantation.

This study aimed to supplement current literature on the safety and efficacy of kidney transplantation in patients with aortoiliac stenosis. To achieve this, all patients undergoing kidney transplantation in Erasmus Medical Center between January 2010 and December 2020 were enrolled, and propensity score matching was used to minimize confounding factors. Additionally, long-term graft function was investigated to evaluate the impact of stenosis on graft function.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent kidney transplantation in the Erasmus Medical Center between January 2010 and December 2020

Exclusion Criteria:

* Patients who were under 18 years at transplantation
* Patients who underwent combined organ transplantation
* Patients who had no follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent kidney transplantation in the Erasmus Medical Center between January 2010 and December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 655 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yitian Fang, MD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Yitian Fang, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
The data that support this study are not publicly available due to reasons of sensitivity and are available from the principal investigator upon reasonable request.

REFERENCES:
- [Derived] Fang Y, Hamm JJM, den Hartog FPJ, Kimenai HJAN, de Bruin RWF, Minnee RC. Safety and efficacy of kidney transplantation in patients with aortoiliac stenosis: a retrospective cohort study. Int J Surg. 2024 Feb 1;110(2):992-999. doi: 10.1097/JS9.0000000000000926. PMID 38016127

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We initially identified all patients undergoing kidney transplantation in Erasmus Medical Center between January 2010 and December 2020. The exclusion criteria were age less than 18 years when transplanted, combined organ transplantation, or no follow-up data.
Pre-assignment Details: We initially identified 2127 participants. Thirty-six patients were excluded according to the exclusion criteria. In the remaining participants, propensity score matching was performed in a nearest neighbor-matching approach with a maximum caliper of 0.1 in a 1 : 4 ratio to match the baseline characteristics of participants with and without aortoiliac stenosis. The matching parameters included age at transplant, dialysis mode, retransplant, donor type, comorbidities, and smoking status.
Groups:
- No-stenosis Group: After PSM, patients who had no pre-existing aortoiliac stenosis before kidney transplantation.
Period: Overall Study
Arm/Group | No-stenosis Group | TASC A/B Stenosis | TASC C/D Stenosis
Started | 524 | 96 | 35
Completed | 524 | 96 | 35
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Propensity score matching was performed in a nearest neighbor-matching approach with a maximum caliper of 0.1 in a 1 : 4 ratio to match patients in the stenosis group with individuals from the no-stenosis group who shared similar characteristics. The matching parameters included age, dialysis mode, retransplant, donor type, comorbidities, and smoking status.
Groups:
- TASC A/B Stenosis Group: Patients who had TASC A/B aortoiliac stenosis before kidney transplantation.
- TASC C/D Stenosis Group: Patients who had TASC C/D aortoiliac stenosis before kidney transplantation.
- Total: Total of all reporting groups
Arm/Group | No-stenosis Group | TASC A/B Stenosis Group | TASC C/D Stenosis Group | Total
Number analyzed (Participants) | 524 | 96 | 35 | 655
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [59 to 71] | 66 [60 to 70] | 63 [59 to 69] | 66 [60 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 34 | 10 | 213
  Male | 355 | 62 | 25 | 442
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 28 [24 to 31] | 27 [24 to 32] | 28 [23 to 31] | 28 [24 to 32]
Type of Dialysis [Count of Participants; unit: Participants]
  Pre-emptive | 120 | 24 | 5 | 149
  Hemodialysis | 297 | 52 | 22 | 371
  Peritoneal Dialysis | 69 | 12 | 5 | 86
  Combined Modality | 38 | 8 | 3 | 49
Duration of Dialysis [Median (Inter-Quartile Range); unit: months] | 22 [11 to 36] | 22 [15 to 37] | 26 [15 to 38] | 22 [12 to 38]
Retransplant [Count of Participants; unit: Participants] | 87 | 15 | 6 | 108
Donor Type [Count of Participants; unit: Participants]
  Living Donor | 290 | 55 | 15 | 360
  DBD | 87 | 15 | 6 | 108
  DCD | 147 | 26 | 14 | 187
Smoking Status [Count of Participants; unit: Participants]
  Never Smoker | 150 | 25 | 13 | 188
  Former Smoker | 261 | 50 | 15 | 326
  Current Smoker | 113 | 21 | 7 | 141

OUTCOME MEASURES:

1. Primary Outcome: Patient Survival
Description: Patient survival was calculated based on all-cause death from the date of kidney transplantation till the end of follow-up (January, 2023), assessed up to 10 years.
Time Frame: From the date of kidney transplantation till death or data cut-off, whichever came first, assessed up to 10 years.
Measure: Count of Participants; unit: Participants
Arm/Group | No-stenosis Group | TASC A/B Stenosis | TASC C/D Stenosis
Number analyzed (Participants) | 524 | 96 | 35
Participants | 322 | 48 | 6

2. Secondary Outcome: Death-censored Graft Survival
Description: Death-censored graft survival was calculated based on death-censored graft failure, from the date of kidney transplantation till death or data cut-off, whichever came first, assessed up to 10 years.
Time Frame: From the date of kidney transplantation till death or data cut-off, whichever came first, assessed up to 10 years.
Measure: Count of Participants; unit: Participants
Arm/Group | No-stenosis Group | TASC A/B Stenosis Group | TASC C/D Stenosis Group
Number analyzed (Participants) | 524 | 96 | 35
Participants | 443 | 80 | 26

3. Secondary Outcome: Graft Function
Description: Estimated glomerular filtration rate (eGFR) was calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation at every post transplant year up to 10 years.
Time Frame: From the date of kidney transplantation till death or data cut-off, whichever came first, assessed up to 10 years.
Population: The discrepancy in the number of participants analyzed in one or more rows compared to the overall number of participants was due to attrition from graft failure or patient death over time.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73m2
Arm/Group | No-stenosis Group | TASC A/B Stenosis Group | TASC C/D Stenosis Group
Number analyzed (Participants) | 476 | 81 | 28
mL/min/1.73m2
  1 year posttransplant | 46 [35 to 59] | 51 [40 to 61] | 46 [35 to 54]
  2 years posttransplant: number analyzed (Participants) | 437 | 73 | 22
  2 years posttransplant | 46 [35 to 59] | 50 [37 to 63] | 42 [30 to 52]
  3 years posttransplant: number analyzed (Participants) | 380 | 60 | 17
  3 years posttransplant | 47 [34 to 61] | 47 [33 to 61] | 40 [35 to 45]
  4 years posttransplant: number analyzed (Participants) | 303 | 47 | 15
  4 years posttransplant | 48 [35 to 62] | 41 [32 to 59] | 42 [29 to 50]
  5 years posttransplant: number analyzed (Participants) | 242 | 39 | 14
  5 years posttransplant | 48 [36 to 61] | 40 [28 to 59] | 38 [33 to 48]
  6 years posttransplant: number analyzed (Participants) | 183 | 31 | 13
  6 years posttransplant | 47 [35 to 62] | 46 [30 to 60] | 46 [31 to 49]
  7 years posttransplant: number analyzed (Participants) | 122 | 28 | 11
  7 years posttransplant | 47 [34 to 65] | 45 [26 to 56] | 40 [30 to 47]
  8 years posttransplant: number analyzed (Participants) | 93 | 18 | 3
  8 years posttransplant | 46 [32 to 64] | 50 [39 to 58] | 47 [44 to 57]
  9 years posttransplant: number analyzed (Participants) | 75 | 13 | 3
  9 years posttransplant | 46 [33 to 62] | 46 [40 to 55] | 50 [49 to 58]
  10 years posttransplant: number analyzed (Participants) | 51 | 4 | 3
  10 years posttransplant | 50 [30 to 61] | 35 [25 to 43] | 48 [40 to 59]

ADVERSE EVENTS:
Time Frame: The time frame for adverse event is from the date of kidney transplantation till death or data cut-off, whichever came first, assessed up to 10 years.
Arm/Group | No-stenosis Group | TASC A/B Stenosis | TASC C/D Stenosis
All-Cause Mortality (participants affected / at risk) | 202/524 | 48/96 | 29/35
Serious Adverse Events (participants affected / at risk) | 0/524 | 0/96 | 0/35
Other Adverse Events (participants affected / at risk) | 0/524 | 0/96 | 0/35

LIMITATIONS AND CAVEATS:
Firstly, there is a guarantee for selection bias in patients with the most severe aortoiliac stenosis, as these patients might be rejected for kidney transplantation and would not be included in the study. Secondly, the study's single-center design could introduce institutional-speciﬁc practices that may not be universally applicable. Lastly, details of stenosis proximal or distal to the transplanted kidney were unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT06020534/Prot_SAP_000.pdf